CLINICAL TRIAL: NCT05709444
Title: A Phase IIb, Multicenter, Open-Label, Prospective Study of Bremelanotide in Diabetic Kidney Disease to Assess the Efficacy in Reducing Urinary Protein and Maintaining Podocyte Density and Function
Brief Title: A Phase IIb, Multicenter, Open-Label, Prospective Study of Bremelanotide in Diabetic Kidney Disease
Acronym: BREAKOUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT-701
Record Dates: First submitted 2023-01-06; First posted 2023-02-02 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-12

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases | interventions — bremelanotide; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, open-label trial to assess the efficacy of melanocortin receptor agonist bremelanotide (BMT) when administered with RAAS inhibition therapy after six months in subjects with Type II diabetic nephropathy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subcutaneous Bremelanotide (Experimental): BMT sterile aqueous solution for injection provided as a prefilled syringe, administered by subcutaneous (SQ) injection into the abdomen.
  Interventions: Drug: Bremelanotide; Drug: RAAS inhibition therapy

INTERVENTIONS:
Drug: Bremelanotide — Bremelanotide is a cyclic, heptapeptide analog of the endogenous peptide alpha melanocortin stimulating hormone (αMSH).
  Other Names: Bremelanotide acetate
Drug: RAAS inhibition therapy — RAS-acting agents are medicines acting on a hormone system that helps to control blood pressure and the amount of fluid in the body.
  Other Names: Angiotensin-converting enzyme (ACE) inhibitors; Angiotensin II receptor blockers (ARBs)

SUMMARY:
This is a prospective, open-label trial to assess the efficacy of melanocortin receptor agonist bremelanotide (BMT) when administered with RAAS inhibition therapy after six months in subjects with Type II diabetic nephropathy. After six months of therapy, all subjects will remain in trial for further assessment and undergo a diagnostic renal biopsy to assess the effect of melanocortin therapy on diabetic histopathology at 12 months.

DETAILED DESCRIPTION:
A total of 45 subjects with biopsy-proven Type II diabetic nephropathy and >1000 mg/gm UP/Cr ratio will be enrolled to receive BMT therapy in addition to their maximum tolerated RAAS inhibition therapy for six months. The subjects' historical medical and laboratory data collected at four timepoints, approximately 24, 18, 12, and 6 months prior to Day 0, will be reviewed and recorded to be used as baseline values.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 years and 80 years, inclusive, willing, and able to understand the risks of the trial and consents to trial conduct documented by the signing of the trial informed consent form.
2. Have a diagnosis of Type II diabetes mellitus in a controlled state (defined as Hemoglobin A1c (HgbA1c) ≤ 10%). Note: Efforts will be made to enroll subjects with known diabetic retinopathy and diabetic peripheral neuropathy to examine the potential benefits of melanocortin receptor activation outside kidney disorders.
3. Have a BMI ≤ 45 kg/m^2 at screening.
4. Have a diagnosis of Stage I, II, or III diabetic nephropathy, confirmed by renal biopsy within 5 years of Screening.
5. Have been on a stable dose of oral diabetic agents or insulin injections for ≥3 months prior to enrollment. Sliding scale dose of insulin based on blood sugar readings is acceptable as long as the type of insulin has remained stable.
6. Be on a stable, maximum tolerated dose (as determined by the Investigator) of an angiotensin-converting enzyme (ACE) or angiotensin-receptor blockers (ARB) as primary antihypertensive therapy (blood pressure of <140/90 at screening).

   Note: If the blood pressure is >140/90 at screening it can be repeated twice and if it is <140/90 upon repeat the subject is eligible for study enrollment.

   Note: The addition or dose modification of ACE-ARB agents after consent is not allowed unless for a safety reason and in consultation with the Medical Monitor prior to adding or modifying.

   Note: Subjects requiring additional medications to achieve the target blood pressure will use antihypertensive agents that have neutral effects on urinary proteinuria (e.g., Hydralazine or long-acting Dihydropyridine calcium channel blockers, etc.).
7. Any subject taking Finerenone, Spironolactone, Eplerenone or any other mineralocorticoid receptor antagonists (MRAs), SGLT inhibitors, and non-dihydropyridine channel blockers (e.g., Diltiazem and Verapamil) must have been on a stable dose for ≥3 months prior to enrollment.

   Note: The addition or dose modification of these agents after consent is not allowed unless for a safety reason and in consultation with the Medical Monitor prior to adding or modifying.
8. Any subject taking a medication that the Investigator believes could alter urinary protein or eGFR must agree to maintain a stable dose throughout the study period, including SGLT2 inhibitors.

   Note: Insulin and other diabetic agents can be adjusted for glycemic control.
9. Have an eGFR by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula ≥20ml/min/1.73m^2, at screening.
10. At screening, two first morning urinary voids obtained with an average UP/Cr ratio of >1,000 mg/gm. If the FMV values are not met, a 24-hour urine collection of protein can be completed and must average UP/Cr ratio of > 1,000 mg/gm for study inclusion.
11. For female subjects:

    1. Women of childbearing potential (WOCBP) must agree to abstain from heterosexual intercourse or use a highly effective contraceptive(s) (with a failure rate of <1% per year), as described in the protocol, during the treatment and follow-up and for at least 90 days after the last dose of BMT. Female Subjects must agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this 90-day period. Hormonal-based contraception is to be employed for a minimum of 28 days prior to Day 0. The Investigator should evaluate the effectiveness of the contraception method in relation to the dose of the investigational product. Note: Oral hormonal contraceptives should be combined estrogen and progesterone. If a progesterone-only oral contraceptive is used, then a second method of birth control should be used as well.
    2. Alternatively, a female of non-childbearing potential is defined as:

    i. Age ≥ 50 years, no menses for at least one year, per subject self-report. ii. Documented hysterectomy, bilateral tubal ligation, or bilateral oophorectomy.
12. For male subjects:

    1. Agree to abstain from heterosexual intercourse or use double barrier protection with condom and spermicide with any WOCBP sexual partner from screening and continuing for at least 30 days after the administration of BMT. Male subjects must also agree not to donate sperm during these 30 days.
    2. Alternatively, documented sterilization confirmed by the absence of sperm in the ejaculate or ≥ one-year post-operative from vasectomy.

Exclusion Criteria

Subjects will be excluded from the trial if they meet any of the following criteria:

1. Females who are pregnant or breastfeeding or plan to become pregnant or donate ova during the trial or 30 days after trial participation.
2. Has a known allergy or intolerance to AECI, ARB, or Melanocortin peptides.
3. Patients with a positive Serum Antigen/Antibody Hepatitis Panel (Hep B and C) and HIV antibody test Human Immunodeficiency Virus (HIV) antibody.

   Note: Patient with positive hepatitis C antibody but negative PCR test for active Hepatitis C viral shedding will be allowed to participate in the study. Patients with a positive Hepatitis B surface antigen antibody or core antigen antibody will be allowed to participate in the study. Patients with circulating hepatitis B surface antigen or have a positive PCR test for active hepatitis B virus will NOT be allowed to participate in the study.
4. Patients with a known active history of alcohol dependence and/or drug use (with Cannabis exception) will be excluded from the study.
5. Has significant medical illnesses that cannot be adequately controlled with appropriate therapy and may obscure toxicity, dangerously alter drug metabolism, or compromise the subject's ability to participate in the trial, as determined by the Investigator.
6. Has current or prior receipt of bremelanotide therapy within the past year.
7. Has used cyclosporine A, adrenocorticotropic hormones, long-term corticosteroids (> 20 mg qd or its equivalent for > 3 months), or cytotoxic agents within the past 3 months.
8. Has a known positive ANA, or Anti-ds-DNA serology and considered by the site principal investigator to have active lupus will NOT be allowed to participate in the study. Patients with a positive RPR but a negative FTA test will be allowed to participate in the study. Patients with a positive Anti-PR3 or Anti-MPO antibody test and thought to have a clinical presentation consistent with ANCA vasculitis will NOT be allowed to participate in the study.
9. Has a solitary kidney (acute kidney injury "AKI" risk) or is on dialysis.
10. Has compromising heart failure or other cardiomyopathies in the opinion of the site Investigator.
11. Has a known history of hyperosmolar states (requiring hospitalization within two months of screening), non-diabetic glomerular disease (with the exclusion of hypertensive glomerulopathy), AKI (requiring renal replacement therapy within two months of screening), kidney transplant, cancer (within 2 years of screening with the exception of non-melanoma skin cancer).
12. Has symptomatic and clinically significant hypotension or dehydration, as determined by the Investigator.
13. Has taken any experimental drug or therapy within 28 days / 5 half-lives of trial treatment or concurrently participating in another clinical trial.
14. Has a history of clinically significant bradycardia and/or a heart rate less than 50 bpm at screening.
15. Plan for blood donations during the study and within 30 days following completion of or early discontinuation from the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of 0.5 mg subcutaneous BMT (given twice a day), used in combination with a subject's maximum tolerated dose of RAAS inhibition therapy, reduces urinary protein by 50% from baseline UP/Cr levels. | Baseline to after six months of combined therapy (RAAS inhibition therapy plus BMT).
  Proportion of subjects with Type II diabetic nephropathy who achieve a 50% reduction in their urine protein Cr (UP/Cr) ratio after six months of combined therapy (RAAS inhibition therapy plus BMT). Inhibition therapy to reduce urinary protein and maintain podocyte density and functions in subjects with Type II diabetic nephropathy after six months.
To determine the incidence of overall adverse events, related adverse events, a composite of adverse events of special interest, serious adverse events, and the incidence of BMT discontinuation. | Baseline to after six months of combined therapy (RAAS inhibition therapy plus BMT).
  Proportion of subjects with Type II diabetic nephropathy who achieve a 50% reduction in their urine protein Cr (UP/Cr) ratio after six months of combined therapy (RAAS inhibition therapy plus BMT) to determine the incidence of adverse events, related adverse events, adverse events of special interest, serious adverse events and BMT discontinuation.

SECONDARY OUTCOMES:
To evaluate the percentage of patients receiving SQ BMT in combination with RAAS inhibition to achieve a complete remission defined as a UP/Cr ratio of ≤ 500 mg/gm at 6 months. | < 500 mg/gm at 6 months.
  Clinical Remission: Proportion of subjects that achieve a reduction in UP/Cr ratios of ≤ 500 mg/gm at 6 months.
To evaluate the percentage of patients receiving SQ BMT in combination with RAAS inhibition to achieve partial remission defined as a UP/Cr ratio of ≥ 50% reduction from baseline UP/Cr at 6 months. | ≥ 50% reduction from baseline UP/Cr at 6 months.
  Partial Remission: Proportion of subjects that achieve a reduction in UP/Cr ratios of ≥ 50% reduction from baseline UP/Cr at 6 months.
To determine the percentage of patients to achieve a clinical response defined as ≥ 30% reduction from BL UP/Cr at 6 months. | ≥ 30% reduction from BL UP/Cr at 6 months.
  Proportion of subjects that achieve a reduction in UP/Cr ratios of ≥ 30% reduction from baseline UP/Cr at 6 months.
To measure the percentage of subjects receiving SQ BMT in combination with RAAS inhibition therapy whose eGFR decreases by less than 5.0 mL/min/1.73m2 from baseline at 6 months. | <5.0mL/min/1.73m^2 from baseline at 6 months.
  Proportion of subjects with Type II diabetic Nephropathy receiving maximally tolerated renin-angiotensin (RAAS) blockade, experiencing a reduction in eGFR of less than 5.0 mL/min/1.73m2 from baseline at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jordan, Study Director — Palatin; James Tumlin, MD, Principal Investigator — Georgia Nephrology Research Institute
Locations (9):
- United States (9):
  - California Institute of Renal Research, Chula Vista, California
  - California Institute of Renal Research DBA - Balboa Research, La Mesa, California
  - Georgia Nephrology, LLC DBA -GA Nephrology Research Institute, Decatur, Georgia
  - Georgia Nephrology, LLC [DBA] GA Nephrology Research Institute, Lawrenceville, Georgia
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Northeast Research Center, LLC, Bethlehem, Pennsylvania
  - Nephrotex Research Group, Dallas, Texas
  - Prolator Clinical Research Center, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No